CLINICAL TRIAL: NCT03013647
Title: Daylight Photodynamic Therapy for Actinic Keratosis and Skin Field Cancerization - Clinical and Histopathological Analysis
Brief Title: Daylight Photodynamic Therapy for Actinic Keratosis and Skin Field Cancerization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, BENI MOREINAS GRINBLAT, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.788.362
Record Dates: First submitted 2016-11-28; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; field cancerization; photodynamic therapy; daylight photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Actinic Keratosis (Other): Twenty patients with multiple thin AK on the face will be treated with Daylight Photodynamic Therapy with methyl aminolevulinate Skin biopsies before and after treatment will be performed in an AK lesion and in a field cancerization area.
  Interventions: Drug: Methyl Aminolevulinate

INTERVENTIONS:
Drug: Methyl Aminolevulinate — Patients will be treated with Daylight Photodynamic therapy, following these steps:
  1. mild curettage of the AK lesions
  2. application of a chemical sunscreen SPF 30
  3. application of methyl aminolevulinate cream (Metvix R, Galderma Laboratories)
  4. exposition to daylight, for 120 minutes
  5. cleaning of the face
  Other Names: Metvix

SUMMARY:
Twenty patients with multiple actinic keratosis on the face will be enrolled in the study and will be treated with Daylight Photodynamic therapy.

Before and after skin biopsies will be performed, for histological and immunohistochemical analysis.

DETAILED DESCRIPTION:
Twenty patients with multiple thin actinic keratosis (AK) on the face will be included in the study. They will be informed of the procedure in detail and sign a consent form.

Digital photographs will be done in a standardized way. Prior to treatment, all patients will undergo 2 skin biopsies under local anesthesia and with a 2 mm punch biopsy. One biopsy will be done over an AK lesion and the other in an area with no apparent AK (field cancerization).

The patients will be treated with Daylight Photodynamic Therapy, following these steps:

1. mild curettage of the AK lesions
2. application of a chemical sunscreen with sun protection factor (SPF) 30
3. application of methyl Aminolevulinate cream (Metvix R, Galderma Laboratories)
4. exposition to daylight, for 120 minutes
5. cleaning of the face

Three months after treatment, two new skin biopsies will be collected, 1cm away from the initial biopsies. On the same date, new photographs will be made following the same standards as pre-treatment photographs.

ELIGIBILITY:
Inclusion Criteria:

-multiple (at least five) actinic keratosis on the face, grades I and II

Exclusion Criteria:

* phototypes IV, V and VI
* patients treated for actinic keratosis up to 6 months before
* history of allergy to methyl aminolevulinate
* history of photoallergy
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 3 months after treatment
  Counting of Actinic keratosis

SECONDARY OUTCOMES:
Histological changes | 3 months after treatment
  Histopathologic analysis in skin biopsies
immunochemistry changes | 3 months after treatment
  immunochemistry analysis in skin biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Cyro Festa, md, Study Chair — Hospital das Clinicas da USP
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fargnoli MC, Piccioni A, Neri L, Tambone S, Pellegrini C, Peris K. Long-term efficacy and safety of daylight photodynamic therapy with methyl amninolevulinate for actinic keratosis of the face and scalp. Eur J Dermatol. 2017 Feb 1;27(1):89-91. doi: 10.1684/ejd.2016.2882. No abstract available. PMID 27748261
- [Background] Grinblat B, Galimberti G, Pantoja G, Sanclemente G, Lopez M, Alcala D, Torezan L, Kerob D, Pascual T, Chouela E. Feasibility of daylight-mediated photodynamic therapy for actinic keratosis throughout the year in Central and South America: a meteorological study. Int J Dermatol. 2016 Sep;55(9):e488-93. doi: 10.1111/ijd.13256. Epub 2016 Apr 7. PMID 27061814
- [Background] Philipp-Dormston WG, Sanclemente G, Torezan L, Tretti Clementoni M, Le Pillouer-Prost A, Cartier H, Szeimies RM, Bjerring P. Daylight photodynamic therapy with MAL cream for large-scale photodamaged skin based on the concept of 'actinic field damage': recommendations of an international expert group. J Eur Acad Dermatol Venereol. 2016 Jan;30(1):8-15. doi: 10.1111/jdv.13327. Epub 2015 Nov 9. PMID 26552049
- [Background] Grinblat B, Galimberti G, Chouela E, Sanclemente G, Lopez M, Alcala D, Torezan L, Pantoja G. Daylight-mediated photodynamic therapy for actinic damage in Latin America: consensus recommendations. Photodermatol Photoimmunol Photomed. 2016 Mar;32(2):81-7. doi: 10.1111/phpp.12221. Epub 2015 Dec 9. PMID 26541910